CLINICAL TRIAL: NCT05722379
Title: Left Bundle Branch Pacing Versus Right Ventricular Pacing in Patients With Atrioventricular Block: an Observational Cohort Study
Brief Title: Left Bundle Branch Pacing Versus Right Ventricular Pacing in Patients With Atrioventricular Block
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhongxiu Chen, Dr, cardiology department, principal investigator, West China Hospital
Other Study IDs: WestChinaH-LBBP-001
Record Dates: First submitted 2023-01-31; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: AVB - Atrioventricular Block
Keywords: Left bundle branch pacing; Right ventricular pacing; Mortality; Systolic dyssynchrony
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- high-grade AVB patients undergoing permanent pacemaker implantations
  Interventions: Procedure: left bundle branch pacing (LBBP); Procedure: Right ventricular pacing (RVP)

INTERVENTIONS:
Procedure: left bundle branch pacing (LBBP) — After recording the His potential, the 3830-69 lead (Medtronic Inc., Minneapolis, MN USA) was sent 1-2 cm forward and downward to find the insertion point of the right side of intra-ventricular septum combined with the pre-rotation impedance and ECG changes. Ultimately, the tip was perpendicularly straightforward posited against the septum to the left septal side .
Procedure: Right ventricular pacing (RVP) — Right ventricular pacing (RVP) is the standard treatment for patients with continuous ventricular pacing needs.

SUMMARY:
Although emerging evidence demonstrated that left bundle branch pacing (LBBP) is a promising alternative for patients with either a bradycardia or a heart failure pacing indication. However, a direct comparison of the safety, efficacy and LV systolic synchrony between LBBP and RVP regimens was rare. In this study, the investigators aim to conduct a comparison of the safety and effectiveness performance between these two pacing methods for patients with atrioventricular block (AVB). The investigators focused on AVB patients undergoing permanent pacemaker implantations from the 1st of January 2018 to the 18th of November 2021 at West China Hospital.

DETAILED DESCRIPTION:
Right ventricular pacing (RVP) is the standard treatment for patients with continuous ventricular pacing needs. However, clinical studies have shown that RVP can cause electrical and mechanical dyssynchrony of the left ventricle and increase the risks of cardiac insufficiency, atrial fibrillation (AF) and death. Although emerging evidence demonstrated that left bundle branch pacing (LBBP) is a promising alternative for patients with either a bradycardia or a heart failure pacing indication. However, a direct comparison of the safety, efficacy and LV systolic synchrony between LBBP and RVP regimens was rare. In this study, the investigators aim to conduct a comparison of the safety and effectiveness performance between these two pacing methods for patients with atrioventricular block (AVB). The investigators focused on AVB patients undergoing permanent pacemaker implantations from the 1st of January 2018 to the 18th of November 2021 at West China Hospital.

ELIGIBILITY:
Inclusion Criteria:

* included consecutively high-grade AVB patients undergoing permanent pacemaker implantations from the 1 s t of January 2018 to the 18 thof November 2021 at West China Hospital

Exclusion Criteria:

* patients with pacemaker replacements were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutively high-grade AVB patients undergoing permanent pacemaker implantations from the 1 s t of January 2018 to the 18 thof November 2021 at West China Hospital
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
composed of all-cause mortality, lead failure and heart failure hospitalization (HFH) during the follow-ups | through study completion, an average of 2.45 year
  composed of all-cause mortality, lead failure and heart failure hospitalization (HFH) during the follow-ups
Lead failure | through study completion, an average of 2.45 year
  reintervention for increased pacing thresholds, lead dislocation or ventricular perforation after the initial implantation procedure
HFH | through study completion, an average of 2.45 year
  HFH was defined as the admission to hospital for >24 hours with worsening symptoms and signs of heart failure and requiring one or more intravenous diuretics or intravenous inotropic medications

SECONDARY OUTCOMES:
peri-procedure complication | through study completion, an average of 2.45 year
  included pericardial tamponade and pneumothorax
cardiac death | through study completion, an average of 2.45 year
  documented arrhythmogenic death, an unexpected presumed pulseles condition with the absence of an obvious noncardiac explanation, or a death due to congestive cardiac failure or structural heart disease
recurrent unexplained syncope | through study completion, an average of 2.45 year
  recurrent unexplained syncope

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Sichuan, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen Z, Xu Y, Jiang L, Zhang R, Zhao H, Liu R, Zhang L, Li Y, Liu X. Left Bundle Branch Area Pacing versus Right Ventricular Pacing in Patients with Atrioventricular Block: An Observational Cohort Study. Cardiovasc Ther. 2023 Aug 21;2023:6659048. doi: 10.1155/2023/6659048. eCollection 2023. PMID 37645544